CLINICAL TRIAL: NCT00226278
Title: Prospective, Double Blind, Randomized, Placebo-Controlled Dose Finding Study of the Efficacy and Safety of 2 Target Doses of Org 34517 Used as Adjunct"
Brief Title: Safety Study of ORG 34517 for Major Depression With Psychotic Features
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: James H. Kocsis, MD, Weill Cornell Medical College
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 28130
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Major Depressive Disorder; Psychotic Disorders
MeSH Terms: conditions — Depressive Disorder, Major; Psychotic Disorders | interventions — Org 34517

INTERVENTIONS:
Drug: ORG 34517

SUMMARY:
Patients suffering from Major Depressive Disorder with Psychotic features who have received no changes in their medications in the previous two weeks will receive "usual" treatment of antidepressants, antipsychotics and/or mood stabilizers and adjunct therapy using ORG34517. The patient will be hospitalized for up to two weeks to monitor their medications and progress and will return to the site for periodic assessments.

ELIGIBILITY:
Inclusion Criteria:

* provide voluntary written informed consent for trial participation after the scope and nature of the investigation have been explained to them, and before starting any trial related activities
* be able to speak, read, understand, respond to questions and follow instructions in English
* have a DSM-IV severe depressive episode with psychotic features, as diagnosed by the MINI for single or recurrent episodes
* have a score on PANSS item "Delusions" AND/OR "Hallucinatory behavior" of at least 4 at screening and baseline
* have a PANSS Positive Scale score of at least 16 at screening and baseline
* have a total score of at least 18 on teh HAMD 17 item scale at Screening and Baseline
* be on a stable dose of usual treatment which has to consist of an anti-depressant, an antipsychotic, a mood stabilizer or any combination of these three drug classes
* be 18 up to and including 70 years of age at Screening
* must be willing to be hospitalized for at least 11 days from Screening onwards.

Exclusion Criteria:

* have any other psychiatric diagnosis except MDD
* have a lifetime psychiatric diagnosis of Bipolar Disorder I, schizophrenia or schizoaffective disorders
* are at significant risk of committing suicide
* are currently treated with carbamazepine or valproate
* are currently treated with midazolam
* have been treated with electroconvulsive therapy in the current episode
* are currently treated with more than one antidepressant
* are currently treated with more than one antipsychotic
* are currently treated with more than one mood stabilizer
* have usual treatment started or discontinued in the two weeks before randomization
* have a usual treatment dose change within the week prior to randomization
* have any clinically unstable or uncontrollable renal, hepatic, respiratory, haematological, cardiovascular or cerebrovascular disease that would put the patient at risk of safety or bias assessment efficacy
* have known hypersensitivity reactions to glucocorticoid antagonists
* have any clinically significant abnormal laboratory data
* have any untreated or uncompensated clinically significant endocrine disorder
* have a diagnosis or alcohol and/or drug dependence
* have a confirmed positive result on the drug screening test for any illicit drug except cannabis
* are using hormone replacement therapy at Screening
* require concomitant treatment with corticosteroids
* are subjects diagnosed with Cushing disease
* are women of childbearing potential without adequate contraception
* are women with a positive pregnancy test at screening or baseline or are breastfeeding mothers
* are male subjects with current diagnosis of prostrate hypertrophia or past history of symptoms of prostrate hypertrophia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2004-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Kocsis, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York, United States